CLINICAL TRIAL: NCT02186548
Title: Closed Versus Open Surgical Exposure of Palatally Displaced Canines (PDC); Treatment and Treatment Outcome Including Aspects of Cost-benefit and Patients´Perceptions. A Multicenter Prospective Randomized Clinical Trial
Brief Title: The Impact of Surgical Technique on PDC
Acronym: PDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Sormland County Council, Sweden (Other); Jonkoping County Hospital (Other)
Responsible Party: Principal Investigator, Margitha Björksved, DDS, MSc, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ÖLL-2013/091
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed surgical technique (Active Comparator): After randomization, the PDC:s randomized to this arm, are to undergo closed surgical exposure, which is an intervention to correct the position of PDC:s.
  Interventions: Procedure: Closed surgical technique
- Open surgical technique (Active Comparator): After randomization, the PDC:s randomized to this arm, are to undergo open surgical exposure, which is an intervention to correct the position of PDC:s.
  Interventions: Procedure: Open surgical technique

INTERVENTIONS:
Procedure: Closed surgical technique — * Surgically uncovering of the impacted canine with a mucoperiosteal flap dissected off the bone
  * The bone covering the canine is being removed
  * Attachment with a chain is bonded to the exposed tooth
  * The palatal flap is repositioned and sutured back with the chain above the mucosa. Shortly after the surgery
  * The canine is orthodontically moved beneath the palatal mucosa
  Arms: Closed surgical technique
Procedure: Open surgical technique — * Surgically uncovering of the impacted canine, removing a window of tissue from around the tooth
  * Pack/filling material is applied on the tooth
  * Spontaneous eruption of the palatally impacted canine is allowed expected
  * The canine is orthodontically moved above the mucosa
  Arms: Open surgical technique

SUMMARY:
Permanent canines in the maxilla usually erupt into the mouth at 11-12 years of age. In approximately 2% of the Swedish population they fail to erupt, and are then referred to as impacted. One severe complication of impacted maxillary canines is damage (root resorption) to the roots of adjacent teeth. The root resorption may be so severe that neighboring teeth are lost. If the impaction is detected early (at 9-10 years of age), the recommended treatment is to extract the deciduous canine, to help the permanent canine to resolve its unfavorable position. If there is no improvement of the position of the canine 1 year after the extraction, surgical and orthodontic treatment is indicated. Surgical exposure is followed by orthodontic treatment with fixed appliance for 2 to 3 years to bring the canine into correct position.

Two different main principles of surgical exposure in palatally impacted maxillary permanent canines are the so called closed versus open surgical techniques.

Closed technique involves surgically uncovering of the canine with a mucoperiosteal flap dissected off the bone. The bone covering the canine is being removed and an attachment with a chain is bonded to the tooth. The flap is repositioned and sutured back with the chain above the mucosa. Shortly after the surgery, orthodontic force is applied via the chain. The canine is orthodontically moved beneath the palatal mucosa by forced eruption.

Open technique involves surgically uncovering of the canine, removing a window of tissue around it and placing pack to cover the exposed area. Then the treatment approaches vary depending on whether the attachment with a chain is bonded to the exposed tooth at surgery or if spontaneous eruption of the palatally impacted canine is expected postsurgically. In both alternatives orthodontic force is applied via the chain and the canine is orthodontically moved above the mucosa. These two techniques of surgical exposure of palatally impacted canines seem to be the two routinely used in Sweden.

The purposes of this study are to examine, describe and compare the treatment outcomes in regard to success and duration of treatment, complications, side effects, cost-benefit aspects and patients´ perceptions in closed versus open surgical exposure techniques, in cases with palatally impacted canines.

The objective is to test the null hypothesis that there are no differences in the above outcomes between open or closed surgical exposure of palatally impacted canines.

DETAILED DESCRIPTION:
Methods of exposing canines are today left to the personal choice of the surgeon and orthodontist. According to an unpublished survey among orthodontists in Sweden 2012, 80% of them use the closed technique only, 9% use the open technique only and 11% use both techniques. This result may be compared to a similar survey performed in the UK, where 29% selected a closed surgical technique only, 40% selected an open surgical technique only and the remainder chose combinations of techniques.

Mentioned reasons for preference of the closed technique are less pain and need for analgesics and faster recovery of pain, postsurgically. Some orthodontists that prefer the open exposure technique have experienced more patient related pain or discomfort in the closed exposure technique, in association with activation in orthodontically forced eruption, because the palatally impacted canine is moved beyond the mucoperiosteal flap. There are no previous studies in this aspect, though.

Factors as operation time, total treatment time and periodontal health measurements after surgical exposure and orthodontic forced eruption of impacted canines, have shown heterogeneity in different retrospective studies.

The management of the palatally impacted canines is a multidisciplinary, time consuming treatment, contributing to relatively high society costs, why this study is taking place, trying to clarify some issues in the choice of method and treatment.

Subjects Patients with diagnosis of uni- or bilateral palatally impacted canine/-s planned for surgical exposure are included consecutively at three orthodontic centers of the Public Dental Health Service in the towns of Orebro, Eskilstuna and Jönköping, Sweden.

Procedure At the appointment for treatment information, the orthodontist gives potential study participants and their parents verbal and written information about the trial. The potential study participants and their parents will be allowed at least one week to decide whether to participate in the trial and if they agree to participate, the written consent will be submitted to the orthodontic centre.

After informed consent is obtained, the participants are randomly allocated to 1 of 2 interventions.

A computer generated randomization is undertaken to ensure that there are equal numbers allocated to each intervention. Allocation concealment is held by one individual per centre, not involved with the trial, who will be contacted by the consenting clinician when the patient is going to be referred for surgical exposure. There will be no stratification for age or gender into the two different groups.

If maxillary deciduous canine are present; they are removed at the time of surgical exposure. The two different surgical exposure techniques are described under "Intervention arms".

The patients are given verbal and written postsurgical information.

Verbal pre-/postsurgical information consists of the recommendation of:

* Analgetic (paracetamol first choice) 1 hour before surgery and there after every 6 to 8th hour 2 days post surgically, according to the dosage recommended
* Tooth paste without sodium is recommended when used directly in association with chlorhexidine rinse

Together with the written postsurgical information, a questionnaire is handed out at the surgical clinic to the patients, for assessment of their experience of pain and discomfort in the evening of the day of surgical exposure and one week there after. The postsurgical questionnaire contains questions that are validated. This questionnaire is submitted to the orthodontic centre at the first postsurgical control.

After surgical exposure orthodontic force is applied; in the closed technique group no later than 2 weeks post surgically and in the open technique group when bonding attachment is possible. In both surgical exposure groups orthodontic force is applied to the palatally impacted canine via the chain attached to the bonded attachment on the canine, to a fixed orthodontic appliance.

Questionnaires are handed out to the patients every 3rd month at the orthodontic clinic, to evaluate the patients´ perceptions of pain and discomfort, until the impacted canine is orthodontically positioned in the dental arch. These questionnaires are submitted at the orthodontic clinic the same day, in association with orthodontic appointment. Questionnaire to assess patients´ perceptions of dental anxiety is handed out to the patient before treatment, when the impacted canine has erupted and when active treatment is finished in each surgical exposure group, at the orthodontic centre. Dental anxiety will be evaluated and described according to Cuthbert MI and Melamed BG. The patients are followed until the active orthodontic treatment is finished and an orthodontic retainer is fitted.

Observation schedule and material/registrations:

Before surgical treatment (T0):

* Impression for study cast/ Registrations: sagittal, transversal and vertical relation, crowding and spacing of teeth (measured according to the current clinical routine), maxillary dental development stage according to Björk
* Panoramic radiograph/ Registrations: mesial position of the impacted canine crown, mesial inclination of the canine to the midline, distance to the occlusal line according to Ericson and Kurol
* CBCT (cone beam computed tomography) examination/ Registrations: exact position and follicle size of the impacted canine; crestal bone height in the lateral incisor in the impacted and nonimpacted contra lateral side in the same patient; root resorption in the impacted canine, the incisors and the eventual first premolar in the impacted and nonimpacted contra lateral side in the same patient
* Clinical examination (according to clinical routine)/ Registrations: periodontal pocket depth, gingival bleeding on probing, gingival recession; in the lateral incisor in the impacted and nonimpacted contra lateral side in the same patient
* CFSS-DS (dental anxiety) questionnaire/ Assessment of dental anxiety
* Registration of age, gender, presence of deciduous canine and date of eventual extraction of deciduous canine

The day of surgical exposure (T1):

* A questionnaire (for the first evening and one week after surgical exposure)/ Assessment of experience of pain, discomfort (measured in VAS-scales) and consumption of analgesics one week after surgical exposure
* Measurement and registration of operation duration

Palatally impacted canine erupted; here: when bonding attachment is possible/ approximately ⅓-½ of the clinical crown of the impacted canine is exposed intraorally (T2):

* Measurement and registration of the duration for the canine to erupt into the oral cavity; time between T1 and T2
* Registration of presence, type and number of complications/failures associated with surgical technique
* CFSS-DS questionnaire/ Assessment of dental anxiety

Previously impacted canine positioned in the dental arch; here: canine ligated to .016x.022 nickel titanium/standard steel arch-wire in the .018-appliance system and .019x.025 nickel-titanium/ standard steel arch-wire in the .022-appliance system (T3):

* Registration of presence, type and number of complications/failures associated with orthodontic treatment
* Measurement and registration of duration between T2 and T3

Orthodontic retainer is fitted/ Active treatment finished (T4):

* Impression for study cast/ Registration of sagittal, transversal/ vertical relation, crowding/spacing of teeth (measured according to the current clinical routine)
* Clinical examination(according to clinical routine/ Registration of pocket depth, gingival bleeding on probing, gingival recession in the canine, the lateral incisor and the first premolar in the impacted and nonimpacted contra lateral side in the same patient
* CFSS-DS questionnaire/ Assessment of dental anxiety
* Measurement and registration of duration between T3 and T4

Within 2 months after active treatment is finished (retainer fitted):

• CBCT examination/ Registration of crestal bone height in the canine, the lateral incisor and the first premolar in the impacted and nonimpacted contra lateral side in the same patient; root resorption in the canine, the incisors and the first premolar in the impacted and nonimpacted contra lateral side in the same patient

Between the day of surgical exposure (T1) and the day when the previously impacted canine is positioned in the dental arch; here: canine inligated to .016x.022 nickel titanium/ standard steel arch-wire in the .018-appliance system and .019x.025 nickel-titanium/ standard steel arch-wire in the .022-appliance system (T3):

• A questionnaire is handed out to the patient every 3rd month at orthodontic appointments between T1 and T3/ Assessment of patients´ perceptions of pain and discomfort (measured in VAS-scales) and consumption of analgesics

Ethical aspects The Regional Ethic Board of Uppsala University, Uppsala, Sweden, which follows the guidelines of the Declaration of Helsinki has approved the study. The Radiation Protection Boards of the County Councils of Örebro, Eskilstuna and Jönköping have approved the planned radiographic examinations in the study. Patientdata are processed according to the laws Personuppgiftslagen, PUL, (1998:204) and Patientdatalagen (2008:355). The examinations and treatments used in this trial are the current examinations and treatments of palatally impacted canines in Sweden, which have been practiced during several years. All surgical exposures and orthodontic treatments are performed by specialists in dental pediatrics/ clinicians and specialists in orthodontics, respectively, with many years of surgical experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of uni- or bilateral palatally impacted canine/-s planned for surgical exposure at start of treatment of the impacted canines. In the bilateral impaction cases, the impacted canine in the more severe position according to the criteria (in Zone 2-4) proposed by Ericson and Kurol is included in the trial.
* Dental development stage: maxillary DS2M1 and DS3M2 according to Björk
* Pretreatment mesial position of the impacted canine in Zone 2-4, according to the criteria proposed by Ericson and Kurol, documented in panoramic radiographs.

Exclusion Criteria:

* Diseases affecting the somatic and/or craniofacial growth
* Diseases not compatible with anaesthesia or surgery
* Known neuropsychiatric diagnosis or documented learning disability
* Problem to understand Swedish (patient and parent). Interpreter needed
* Patients older than 16 years of age at the year of start of treatment
* Ongoing orthodontic treatment
* Patients with agenesis of the lateral incisor in the impacted side
* Pretreatment mesial position of the impacted canine in Zone 5, according to the criteria proposed by Ericson and Kurol, documented in panoramic radiographs
* Pretreatment vertical position of the impacted canine above the full length root of the central incisor on the same side, according to Fleming, PS. et al.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2013-06; Primary Completion 2021-01 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Treatment success; the previous impacted canine is positioned in the dental arch | Within 3 years after surgery
  "Positioned in the dental arch"; here meaning that the previous impacted canine has been treated with fixed orthodontic braces and is inligated in .016x.022 nickel titanium/ standard steel arch-wire in a .018- appliance system and .019x.025 nickel-titanium/ standard steel arch-wire in a .022- appliance system.

SECONDARY OUTCOMES:
Duration from surgery until the previous impacted canine has erupted into the mouth | Within 1,5 year from surgery
  "Erupted into the mouth"; here meaning that approximately ⅓-½ of the clinical crown of the impacted canine is exposed intraorally.

OTHER OUTCOMES:
Presence, type and number of complications/failures associated with the operation techniques | Within 1,5 years from surgery
Operation time (hours, minutes) | Within 6 months from allocation
Estimation of total treatment costs | Within 3,5 years from surgery
Patients´perceptions of experienced pain, discomfort and consumption of analgesics. | Within 3 years from surgery
  Patients´perceptions of experienced pain, discomfort and consumption of analgesics is registered in questionnaires at the first evening and one week after surgical exposure and every 3rd month until the impacted canine is positioned in the dental arch.
Presence of dental anxiety (patient) and eventual change in dental anxiety during treatment | Within 3 years from surgery
  A Dental Subscale of the Children´s Fear Survey Schedule, CFSS-DS questionnaire will be handed out to the patients at three times (before start of treatment, after the impacted canine has erupted and when the canine is positioned in the dental arch). Dental anxiety and eventual change in dental anxiety will be described, compared and evaluated compared between the two surgical exposure group and individually.
Dental health comparison between the two groups of different surgical exposure | Within 3,5 years from surgery
  Dental health is measured before start of treatment and when treatment is finished, and compared between the surgical groups and also between the impacted and non impacted side in the individual, here as:
  * Periodontal health measured as pocket depth, bleeding on probing and recession of the gingival margin (clinical routine examination)
  * Crestal bone height and eventual root resorption (cone beam computed tomography)

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Bazargani, DDS, PhD, Study Director — Centrum för specialisttandvård, avdelningen för ortodonti, Klostergatan 26, 703 61 Örebro. Tel: 0046-019-6024050
Locations (3):
- Sweden (3):
  - Tandregleringen, Kungsgatan. 21A, Eskilstuna
  - Odontologiska institutionen, avdelningen för ortodonti, Hermansvägen 5, Jönköping
  - Centrum för specialisttandvård, avdelningen för ortodonti, Klostergatan 26, Örebro

REFERENCES:
- [Background] Parkin N, Benson PE, Thind B, Shah A. Open versus closed surgical exposure of canine teeth that are displaced in the roof of the mouth. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006966. doi: 10.1002/14651858.CD006966.pub2. PMID 18843740
- [Background] Spencer HR, Ramsey R, Ponduri S, Brennan PA. Exposure of unerupted palatal canines: a survey of current practice in the United Kingdom, and experience of a gingival-sparing procedure. Br J Oral Maxillofac Surg. 2010 Dec;48(8):641-4. doi: 10.1016/j.bjoms.2009.08.032. Epub 2009 Nov 3. PMID 19889488
- [Background] Parkin NA, Deery C, Smith AM, Tinsley D, Sandler J, Benson PE. No difference in surgical outcomes between open and closed exposure of palatally displaced maxillary canines. J Oral Maxillofac Surg. 2012 Sep;70(9):2026-34. doi: 10.1016/j.joms.2012.02.028. Epub 2012 Jun 6. PMID 22677328
- [Background] Gharaibeh TM, Al-Nimri KS. Postoperative pain after surgical exposure of palatally impacted canines: closed-eruption versus open-eruption, a prospective randomized study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Sep;106(3):339-42. doi: 10.1016/j.tripleo.2007.12.025. Epub 2008 Jun 11. PMID 18547839
- [Background] Pearson MH, Robinson SN, Reed R, Birnie DJ, Zaki GA. Management of palatally impacted canines: the findings of a collaborative study. Eur J Orthod. 1997 Oct;19(5):511-5. doi: 10.1093/ejo/19.5.511. PMID 9386337
- [Background] Caprioglio A, Vanni A, Bolamperti L. Long-term periodontal response to orthodontic treatment of palatally impacted maxillary canines. Eur J Orthod. 2013 Jun;35(3):323-8. doi: 10.1093/ejo/cjs020. Epub 2012 Apr 24. PMID 22531665
- [Background] Fleming PS, Scott P, Heidari N, Dibiase AT. Influence of radiographic position of ectopic canines on the duration of orthodontic treatment. Angle Orthod. 2009 May;79(3):442-6. doi: 10.2319/042708-238.1. PMID 19413390
- [Background] Iramaneerat S, Cunningham SJ, Horrocks EN. The effect of two alternative methods of canine exposure upon subsequent duration of orthodontic treatment. Int J Paediatr Dent. 1998 Jun;8(2):123-9. doi: 10.1046/j.1365-263x.1998.00075.x. PMID 9728097
- [Background] Schmidt AD, Kokich VG. Periodontal response to early uncovering, autonomous eruption, and orthodontic alignment of palatally impacted maxillary canines. Am J Orthod Dentofacial Orthop. 2007 Apr;131(4):449-55. doi: 10.1016/j.ajodo.2006.04.028. PMID 17418710
- [Background] Woloshyn H, Artun J, Kennedy DB, Joondeph DR. Pulpal and periodontal reactions to orthodontic alignment of palatally impacted canines. Angle Orthod. 1994;64(4):257-64. doi: 10.1043/0003-3219(1994)0642.0.CO;2. PMID 7978520
- [Background] Zasciurinskiene E, Bjerklin K, Smailiene D, Sidlauskas A, Puisys A. Initial vertical and horizontal position of palatally impacted maxillary canine and effect on periodontal status following surgical-orthodontic treatment. Angle Orthod. 2008 Mar;78(2):275-80. doi: 10.2319/010907-8.1. PMID 18251594
- [Background] Becker A, Kohavi D, Zilberman Y. Periodontal status following the alignment of palatally impacted canine teeth. Am J Orthod. 1983 Oct;84(4):332-6. doi: 10.1016/s0002-9416(83)90349-4. PMID 6578683
- [Background] Hansson C, Rindler A. Periodontal conditions following surgical and orthodontic treatment of palatally impacted maxillary canines--a follow-up study. Angle Orthod. 1998 Apr;68(2):167-72. doi: 10.1043/0003-3219(1998)0682.3.CO;2. PMID 9564427
- [Background] Stewart JA, Heo G, Glover KE, Williamson PC, Lam EW, Major PW. Factors that relate to treatment duration for patients with palatally impacted maxillary canines. Am J Orthod Dentofacial Orthop. 2001 Mar;119(3):216-25. doi: 10.1067/mod.2001.110989. PMID 11244415
- [Background] Bazargani F, Magnuson A, Dolati A, Lennartsson B. Palatally displaced maxillary canines: factors influencing duration and cost of treatment. Eur J Orthod. 2013 Jun;35(3):310-6. doi: 10.1093/ejo/cjr143. Epub 2012 Jan 24. PMID 22275512
- [Background] Kau CH, Durning P, Richmond S, Miotti FA, Harzer W. Extractions as a form of interception in the developing dentition: a randomized controlled trial. J Orthod. 2004 Jun;31(2):107-14. doi: 10.1179/146531204225020391. PMID 15210926
- [Background] Feldmann I, List T, John MT, Bondemark L. Reliability of a questionnaire assessing experiences of adolescents in orthodontic treatment. Angle Orthod. 2007 Mar;77(2):311-7. doi: 10.2319/0003-3219(2007)077[0311:ROAQAE]2.0.CO;2. PMID 17319767
- [Background] Cuthbert MI, Melamed BG. A screening device: children at risk for dental fears and management problems. ASDC J Dent Child. 1982 Nov-Dec;49(6):432-6. No abstract available. PMID 6960031
- [Background] BJOERK A, KREBS A, SOLOW B. A METHOD FOR EPIDEMIOLOGICAL REGISTRATION OF MALOCCLUSION. Acta Odontol Scand. 1964 Feb;22:27-41. doi: 10.3109/00016356408993963. No abstract available. PMID 14158468
- [Background] Ericson S, Kurol J. Early treatment of palatally erupting maxillary canines by extraction of the primary canines. Eur J Orthod. 1988 Nov;10(4):283-95. doi: 10.1093/ejo/10.4.283. No abstract available. PMID 3208843
- [Derived] Bjorksved M, Ryen L, Lindsten R, Bazargani F. Open and closed surgical exposure of palatally displaced canines: a cost-minimization analysis of a multicentre, randomized controlled trial. Eur J Orthod. 2021 Oct 4;43(5):498-505. doi: 10.1093/ejo/cjab052. PMID 34386824
- [Derived] Bjorksved M, Arnrup K, Bazargani SM, Lund H, Magnusson A, Magnuson A, Lindsten R, Bazargani F. Open vs closed surgical exposure of palatally displaced canines: a comparison of clinical and patient-reported outcomes-a multicentre, randomized controlled trial. Eur J Orthod. 2021 Oct 4;43(5):487-497. doi: 10.1093/ejo/cjab015. PMID 34114630
- [Derived] Bjorksved M, Arnrup K, Lindsten R, Magnusson A, Sundell AL, Gustafsson A, Bazargani F. Closed vs open surgical exposure of palatally displaced canines: surgery time, postoperative complications, and patients' perceptions: a multicentre, randomized, controlled trial. Eur J Orthod. 2018 Nov 30;40(6):626-635. doi: 10.1093/ejo/cjy070. PMID 30321323